CLINICAL TRIAL: NCT04471155
Title: Comparison of Holmium Laser Enucleation Prostatectomy and Open Transvesical Prostatectomy in Large Prostate More Than 80 Grams in Egyptian Men
Brief Title: Comparison of Holmium Laser Enucleation Prostatectomy and Open Transvesical Prostatectomy in Large Prostate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, mohamed alnoomani, mohamed nabil alnoomani, assistant lecturer of urology, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MD/152/2018
Record Dates: First submitted 2020-07-09; First posted 2020-07-15 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Holep (Active Comparator): patient underwent laser prostatectomy
  Interventions: Procedure: Holep
- open prostatectomy (Active Comparator): patient underwent open prostatectomy
  Interventions: Procedure: Holep

INTERVENTIONS:
Procedure: Holep — laser enucleation of the gland versus open enucleation
  Other Names: open prostatectomy

SUMMARY:
comparison of holmium laser enucleation prostatectomy and open prostatectomy regarding safety and efficacy in men with prostate larger than 80 grams

ELIGIBILITY:
Inclusion Criteria:

* American Urological Association Symptom Score of eight or higher,
* Maximum urinary flow rate of 10ml/s or less,
* Post void residual urine volume of 50 ml or more,
* And a total prostate volume of 80 ml or more in transrectal ultrasound (TRUS).

Exclusion Criteria:

* A previous prostate or urethral surgery
* And non-BPH related voiding disorders
* Prostate cancer patients

Min Age: 55 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — only males have prostate
Enrollment: 110 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-22 (Actual)

PRIMARY OUTCOMES:
efficacy by measuring maximum urinary flow rate in millilitre per second | 1 year
  change of maximum urinary flow rate in mililiter per second pre and post opeartive
efficacy in american urological association symptom score | 1 year
  change of american urological association symptom score pre and post operative by scale from 1 to 35
efficacy of evacuation by measuring post-voiding residual urine volume in millilitre | 1 year
  change of post-voiding residual urine volume in millilitre

SECONDARY OUTCOMES:
safety by doing blood picture to asses hemoglobin drop | immediate post-operative
  rate of hemoglobin drop post-operatively by gram per decilitre

CONTACTS AND LOCATIONS:
Locations (1):
- Mohamed Alnoomani, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No